CLINICAL TRIAL: NCT00498186
Title: An Open-label Extension Trial to Determine Safety and Tolerability of Long-term Transdermal Application of Rotigotine in Subjects With Idiopathic Restless Legs Syndrome
Brief Title: Long-term Open-label Trial in Idiopathic Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0710
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2011-10

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Neupro®
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Rotigotine trans-dermal patch
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine transdermal patches once daily:
  2.5cm2 (0.5mg/24 hours) 5cm2 (1mg/24 hours) 10cm2 (2mg/24 hours) 15cm2 (3mg/24 hours) 20cm2 (4mg/24 hours)
  Other Names: Neupro®

SUMMARY:
This is a multi-center, open-label extension trial conducted at the same European sites that participated in trial SP 709 (NCT00243217). The trial is designed to collect long-term safety and tolerability, efficacy correlates, and quality of life data in subjects with idiopathic Restless Leg Syndrome (RLS). The duration of treatment is approximately 5 years. Subject will be up-titrated to their optimal dose (administration of 1 patch per day, 5 different doses and patch sizes).

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the preceding trial SP709 (NCT00243217)

Exclusion Criteria:

* Subject did suffer from a serious adverse event during trial SP709 (NCT00243217) which is ongoing at the end of that trial and is assessed to be related to the study medication by the investigator and/or the Sponsor
* Sleep disturbances
* Further clinically relevant concomitant diseases such as polyneuropathy, akathisia, claudication, varicosis, muscle fasciculation, painful legs and moving toes, or radiculopathy
* Other central nervous diseases
* One psychotic episode since start of study SP709
* Any medical or psychiatric condition, which in the opinion of the investigator can jeopardize or would compromise the subject's ability to participate in this trial
* Clinically relevant cardiac dysfunction and arrhythmias
* The subject has at entry in study SP710, a QTc interval ≥ 500 msec and/or a QTc interval which has increased by ≥ 60 msec as compared to the average baseline (Visit 2) QTc interval of study SP709
* Subject has clinically relevant renal dysfunction (serum creatine ≥ 2.0 mg/dl)
* Subject has clinically relevant hepatic dysfunction (total bilirubin > 2.0 mg/dl or ALT and/or AST greater than two times the upper limit of the reference range
* Subject has a newly diagnosed or relapsing neoplastic disease since the start of study SP709
* Subject has a known hypersensitivity to any components of the trial medication or comparative drugs as stated in this protocol
* Subject needs drugs prohibited in the course of this trial: neuroleptics, bupidine, hypnotics, antidepressants, anxiolytic drugs, anticonvulsive therapy, psychostimulatory drugs, other L-Dopa or dopamine agonist therapy, opioids, benzodiazepines, MAO inhibitors, sedative antihistamines, amphetamines
* Subject is abusing alcohol or drug since start of SP709
* Subject is pregnant or nursing or woman of child-bearing potential who is not surgically sterile, two years postmenopausal, or does not practice two combined methods of contraception, unless sexually abstinent
* Subject pursues shift work or is subject to other continuous non-disease-related life conditions which do not allow regular sleep at night
* Subject has clinically relevant vasculopathies (eg, varix or arteriosclerosis)
* Subject has significant skin hypersensitivity to adhesive or other transdermals or recent unresolved contact dermatitis
* Subject has symptomatic orthostatic hypotension, or a systolic blood pressure (SBP) less tham 105mmHg and/or a drop in SBP of > 20mmHg or a drop of > 10mmHg in diastolic BP (DBP) on standing at baseline visit (Visit 1)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2003-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (24):
- Innsbruck, Austria
- Germany (20):
  - Bamberg
  - Berlin
  - Bielefeld
  - Gelsenkirchen
  - Gera
  - Halle
  - Jena
  - Kassel
  - Köthen
  - Marburg
  - Mittweida
  - München
  - Neubrandenburg
  - Oldenburg
  - Regensburg
  - Schwalmstadt-Treysa
  - Schwerin
  - Tuttlingen
  - Ulm
  - Unterhaching
- Spain (3):
  - Alzira, Valencia
  - Barcelona
  - Madrid

REFERENCES:
- [Result] Oertel WH, Benes H, Garcia-Borreguero D, Geisler P, Hogl B, Trenkwalder C, Tacken I, Schollmayer E, Kohnen R, Stiasny-Kolster K; Rotigotine SP710 Study Group. One year open-label safety and efficacy trial with rotigotine transdermal patch in moderate to severe idiopathic restless legs syndrome. Sleep Med. 2008 Dec;9(8):865-73. doi: 10.1016/j.sleep.2008.04.012. Epub 2008 Aug 26. PMID 18753003
- [Result] Hogl B, Oertel WH, Stiasny-Kolster K, Geisler P, Benes H, Garcia-Borreguero D, Trenkwalder C, Poewe W, Schollmayer E, Kohnen R. Treatment of moderate to severe restless legs syndrome: 2-year safety and efficacy of rotigotine transdermal patch. BMC Neurol. 2010 Sep 28;10:86. doi: 10.1186/1471-2377-10-86. PMID 20920156
- [Result] Oertel W, Trenkwalder C, Benes H, Ferini-Strambi L, Hogl B, Poewe W, Stiasny-Kolster K, Fichtner A, Schollmayer E, Kohnen R, Garcia-Borreguero D; SP710 study group. Long-term safety and efficacy of rotigotine transdermal patch for moderate-to-severe idiopathic restless legs syndrome: a 5-year open-label extension study. Lancet Neurol. 2011 Aug;10(8):710-20. doi: 10.1016/S1474-4422(11)70127-2. Epub 2011 Jun 24. PMID 21705273
- [Derived] Dohin E, Hogl B, Ferini-Strambi L, Schollmayer E, Fichtner A, Bauer L, Garcia-Borreguero D. Safety and efficacy of rotigotine transdermal patch in patients with restless legs syndrome: a post-hoc analysis of patients taking 1 - 3 mg/24 h for up to 5 years. Expert Opin Pharmacother. 2013 Jan;14(1):15-25. doi: 10.1517/14656566.2013.758251. Epub 2012 Dec 21. PMID 23256574
- [Derived] Hogl B, Oertel WH, Schollmayer E, Bauer L. Transdermal rotigotine for the perioperative management of restless legs syndrome. BMC Neurol. 2012 Sep 25;12:106. doi: 10.1186/1471-2377-12-106. PMID 23009552
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 295 subjects belong to the Enrolled Set (ES) and all of them received at least one dose of trial medication, so they all belong to the Safety Set (SS).
Pre-assignment Details: Participant Flow information and Baseline Characteristics belong to the Safety Set (SS).
Period: Overall Study
Arm/Group | Rotigotine
Started | 295
Completed | 122
Not Completed | 173
Not completed — Protocol Violation | 10
Not completed — Lack of Efficacy | 31
Not completed — Adverse Event | 89
Not completed — Unsatisfactory compliance of subject | 12
Not completed — Withdrawal by Subject | 18
Not completed — Lost to Follow-up | 3
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 208
  >=65 years | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 99
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/ m^2] — BMI= weight/height^2
  kg/ m^2 | 26.37 (3.84)
Height [Mean (Standard Deviation); unit: cm] | 167.5 (8.3)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 74.21 (13.19)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event, as Reported Spontaneously by the Subject or Observed by the Investigator, During the 5-year Open-label Extension.
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: Up to five years
Population: Of the 295 subjects who entered the study, 295 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 295
participants | 273

2. Secondary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event During the 5-year Open Label Extension
Description: as for outcome 1
Time Frame: Up to five years
Population: Of the 295 subjects who entered the study, 295 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 295
participants | 93

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the whole trial period up to 5 years from Visit 1 to the Safety Follow- up Visit.
Description: Serious and non- serious Adverse Events (AEs) refer to the Safety Set (SS). The SS includes all subjects who received at least one dose of trial medication.
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 79/295
Other Adverse Events (participants affected / at risk) | 272/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=295)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5)
Angina pectoris (Cardiac disorders) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3)
Blood pressure increased (Investigations) | 1 (2)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Toe deformity (Musculoskeletal and connective tissue disorders) | 4 (4)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Impingement syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (13)
Lumbal spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Polyneuropathy (Nervous system disorders) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Sleep apnoe syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominoplasty (Surgical and medical procedures) | 1 (1)
Bladder operation (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 2 (2)
Limb operation (Surgical and medical procedures) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Angioplasty (Surgical and medical procedures) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=295)
Nausea (Gastrointestinal disorders) | 35 (44)
Application site erythema (General disorders) | 96 (132)
Application site reaction (General disorders) | 74 (90)
Application site pruritus (General disorders) | 54 (71)
Fatigue (General disorders) | 31 (36)
Influenza (Infections and infestations) | 15 (17)
Bronchitis (Infections and infestations) | 20 (26)
Nasopharyngitis (Infections and infestations) | 55 (78)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (50)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 (19)
Headache (Nervous system disorders) | 16 (21)
Dizziness (Nervous system disorders) | 16 (20)
Depression (Psychiatric disorders) | 22 (25)
Insomnia (Psychiatric disorders) | 17 (18)
Sleep disorder (Psychiatric disorders) | 21 (22)
Erythemas (Skin and subcutaneous tissue disorders) | 17 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (16)
Hypertension (Vascular disorders) | 26 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.